CLINICAL TRIAL: NCT00584012
Title: A Study of the Proper Dosage of Lovastatin and Docetaxel for Patients With Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding issues
Sponsor: Susan L Roeder (Other)
Responsible Party: Sponsor-Investigator, Susan L Roeder, Physician, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200311038
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-01

CONDITIONS: Any Cancer; Breast Cancer
Keywords: Any cancer; Breast cancer; Lovastatin; Docetaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — Lovastatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Esclation (Experimental): Determine the maximum tolerated dose (MTD) of escalating doses of lovastatin in combination with docetaxel in patients with any type of solid tumor.
  Interventions: Drug: Lovastatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Lovastatin — Given PO
  Other Names: Mevacor
Drug: Docetaxel — Given IV
  Other Names: Taxotere

SUMMARY:
This purpose of this study is to evaluate the use of two medications, docetaxel and lovastatin to determine the highest dose of lovastatin and docetaxel that can be given safely as well as the safety of combining the two drugs and the effect on the subject's tumor. Subjects can have any cancer.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the maximum tolerated dose (MTD) of lovastatin and docetaxel in patients with various different cancers.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of age
* Performance Status (ECOG) <2
* Peripheral Neuropathy < grade I
* Signed Informed consent
* Hematologic-Inclusion Absolute neutrophil count > 1,500/mm3 Hemoglobin > 8.0 g/dl Platelet count > 100,000/mm3.
* Hepatic-Inclusion Total Bilirubin must be within normal limits.
* Transaminases (SGOT and/or SGPT) may be up to 2.5 x institutional upper limit of normal (ULN) if alkaline phosphatase is < ULN, or alkaline phosphatase may be up to 4 x ULN if transaminases are < ULN.
* Patients may have received prior chemotherapy including treatment with the following agents: anthracycline, platinum, vinorelbine, or other Vinca alkaloids. The patient must have recovered from the side effects of the prior treatment including prior drug-induced peripheral neuropathy.
* Patients who have received prior taxane therapy will be eligible. (However, patients who have progressed within 6 months of receiving docetaxel will be excluded.)
* A minimum of 28 days must have elapsed from the completion of any prior chemotherapy or radiation treatment.
* Patients who are currently receiving bisphosphonates for bone disease will be allowed to enter the trial, however their bone lesions will not be considered assessable for response, but will be assessable for progression.
* Initiation of bisphosphonate treatment during the trial will be discouraged but allowed in the absence of progressive disease. If bisphosphonates are initiated, then bone lesions will be assessed for progression only.

Exclusion Criteria:

* Other serious illnesses, which would limit survival to <2 months, or a psychiatric condition, which would prevent compliance with treatment or informed consent.
* ECOG Performance Status >2
* Anticipated survival < 2 months
* Uncontrolled or severe cardiovascular disease, diabetes, pulmonary disease, or infection, which in the opinion of the treating physician would make this protocol treatment unreasonably hazardous for the patient.
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and considered by their physician to be at less than 30% risk of relapse within one year.
* Patients who have received any investigational agent within the prior 4 weeks.
* Age < 18 as there is no safety data for lovastatin in this age range.
* Patients with a history of severe hypersensitivity reaction to Taxotere® or other drugs formulated with polysorbate 80.
* Patients who have received anticancer endocrine therapy within 4 weeks prior to registration are not eligible.
* Patients currently on daily statin therapy will also be excluded.
* Patients who have progressed within 6 months of receiving docetaxel are not eligible.
* Treatment with the anti-emetic Aprepitant is not allowed.
* Patients who are currently receiving , or have received Herceptin therapy within 4 weeks prior to registration are not eligible.
* Pregnant and/or Nursing. Patients must not be pregnant or nursing at the time of enrollment nor while under the treatment of this protocol. Treatment under this protocol would expose an unborn child to significant risks. Women and men of reproductive potential should agree to use an effective means of birth control.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-04 (Actual); Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Roman, DO, Principal Investigator — University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Esclation: Determine the maximum tolerated dose (MTD) of escalating doses of lovastatin in combination with docetaxel in patients with any type of solid tumor.
  Lovastatin and Docetaxel: Docetaxel (60 mg/m2) will be given on day 0 every three weeks with incrementally increasing doses of lovastatin. Lovastatin will be administered p.o. following a four times a day schedule, for four consecutive days (days -1 to +2) and repeated every three weeks. For purposes of this study, intermittent drug administration, six dose levels, ranging from 2 to 24 mg/kg/day (2, 4, 7, 10, 13, 18, and 24 mg) will be used. Once the maximum tolerated dose (MTD) of lovastatin has been determined, docetaxel will be escalated in a stepwise scheme from 60 to 80 to 100 mg/m2.
Period: Overall Study
Arm/Group | Dose Esclation
Started | 9
Completed | 8
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dose Esclation
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants] — Population: Study was terminated prior to completion.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 6
    >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] — Population: Study terminated prior to completion. Enrollment was halted prematurely and will not resume. Participants are no longer being examined or treated.
  years | 56.1 [29.5 to 71.7]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Study terminated prior to completion. Enrollment was halted prematurely and will not resume. Participants are no longer being examined or treated.
  Participants
    Female | 2
    Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Study terminated prior to completion. Enrollment was halted prematurely and will not resume. Participants are no longer being examined or treated.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 9
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Population: Study terminated prior to completion. Enrollment was halted prematurely and will not resume. Participants are no longer being examined or treated.
  participants
    United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose-limiting Toxicities (DLTs)
Description: To determine the maximum tolerated doses (MTD) of lovastatin and docetaxel in patients with various cancers having solid tumors.
Time Frame: 27 weeks
Population: Study terminated prior to completion. Data not collected. Enrollment was halted prematurely and will not resume. Participants are no longer being examined or treated.
Arm/Group | Dose Esclation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Dose Esclation
All-Cause Mortality (participants affected / at risk) | 4/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Esclation (N=9)
Cardiovascular (Arrhythmia) (Cardiac disorders) | 1 (1)
Infection without neutropenia (Infections and infestations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Kidney Stone (Renal and urinary disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Esclation (N=9)
Hypokalemia (Metabolism and nutrition disorders) | 6 (6)
Thrombocytopenia (Skin and subcutaneous tissue disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Indigestion (Gastrointestinal disorders) | 1 (1)
Amylase (Metabolism and nutrition disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 7 (7)
Headache (General disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Hemmorrhage, nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain, scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (6)
Decreased bicarbonate (Metabolism and nutrition disorders) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Anemia (Metabolism and nutrition disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Abdominal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Vomitting (Gastrointestinal disorders) | 4 (6)
Pain, shoulder (Musculoskeletal and connective tissue disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Flushing, face (Skin and subcutaneous tissue disorders) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Fever (General disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Infection with normal ANC (Infections and infestations) | 1 (1)
Mucositis (Gastrointestinal disorders) | 4 (4)
Occular/visual, peripheral light pulsing (Eye disorders) | 1 (1)
Elevated CPK (Metabolism and nutrition disorders) | 1 (1)
Elevated ALT (Metabolism and nutrition disorders) | 2 (2)
Elevated AST (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Hepatobiliary disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Dyspenea on exertion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Abdominal pain, cramps (Gastrointestinal disorders) | 1 (1)
Neutropenia (General disorders) | 1 (1)
Pain, ankle (Musculoskeletal and connective tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Decreased WBC (Blood and lymphatic system disorders) | 4 (5)
Edema (Cardiac disorders) | 5 (8)
Hypersensitivity reaction (Immune system disorders) | 2 (2) — Back pain, chest pain
Pain/tenderness, periorbital region (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain/cramping, leg (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain, hands (Musculoskeletal and connective tissue disorders) | 3 (3)
Hypercholesterolemia (Metabolism and nutrition disorders) | 2 (2)
Pain, oral cavity (General disorders) | 1 (1)
Insomnia (Nervous system disorders) | 2 (2)
Dysgeusia (Gastrointestinal disorders) | 1 (1) — Taste alteration, intermittent
Ataxia (Nervous system disorders) | 1 (1)
Koilonychia (Skin and subcutaneous tissue disorders) | 1 (1) — Fingernail discoloration, thickening
Blurred vision (Eye disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Dyspepsia/heartburn (Gastrointestinal disorders) | 2 (2)
Elevated creatinine (Renal and urinary disorders) | 1 (1)
Elevated Alkaline phosphatase (Hepatobiliary disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Cardiac disorders) | 3 (3)
Mood alteration, depression (Psychiatric disorders) | 2 (2)
Decreased appetite, anorexia (Gastrointestinal disorders) | 2 (2)
Dizziness/lightheadedness (Nervous system disorders) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 1 (2)
Pain, back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, chest (muscular) (Musculoskeletal and connective tissue disorders) | 1 (1)
Decubitus skin breakdown, gluteal folds (Skin and subcutaneous tissue disorders) | 1 (1)
Pain, neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture, iliac wing (Musculoskeletal and connective tissue disorders) | 1 (1)
Fall (Nervous system disorders) | 1 (2)
Weight gain (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Pain, chest/thoracic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash, facial (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, palmar (Skin and subcutaneous tissue disorders) | 1 (1)
UTI (Renal and urinary disorders) | 1 (1)
Joint achiness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastric reflux (Gastrointestinal disorders) | 1 (1)
Urine color change (Renal and urinary disorders) | 1 (1)
Elevated glucose (Metabolism and nutrition disorders) | 1 (1)
Decreased netrophils (Blood and lymphatic system disorders) | 1 (1)
Pain, hip (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study terminated due to funding issues prior to completion. No data were analyzed. Enrollment was halted prematurely and will not resume. Participants are no longer being examined or treated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No